CLINICAL TRIAL: NCT06600724
Title: A Multicenter, Prospective, Randomized Controlled Modified Platform Trial Evaluating PURION Processed Lyophilized Human Amnion/Chorion Membrane (ppLHACM) and Standard of Care Versus Standard of Care Alone in the Treatment of Nonhealing Diabetic Foot Ulcers
Brief Title: Modified Platform Trial Evaluating PpLHACM and SOC Versus SOC Alone in the Treatment of Nonhealing DFUs
Acronym: CAMPAIGN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIMEDX001
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Foot Ulcer Due to Type 2 Diabetes Mellitus; Foot Ulcer, Diabetic; Foot Ulcer
Keywords: Ulcer; Foot Ulcer; Diabetic Foot Ulcer; Foot
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: CAMPAIGN uses a Prospective Modified Platform Multicenter Randomized Controlled Clinical Trial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (Active Comparator): Standard of care will be cleaning, debridement, ulcer moisture balance, and offloading.
  Interventions: Other: Standard of Care
- EPIEFFECT (Experimental): EPIEFFECT® is a PURION processed lyophilized human placental tissue allograft that includes the amnion layer, intermediate layer, and chorion layer of the amniotic membrane. The product is intended for use as a barrier to provide a protective environment in acute and chronic wounds.
  Interventions: Other: EPIEFFECT
- EPIXPRESS (Experimental): EPIXPRESS™ is a PURION processed lyophilized human placental tissue allograft that includes the amnion layer, intermediate layer, and chorion layer of the amniotic membrane. The product is intended for use as a barrier to provide a protective environment in acute and chronic wounds. EPIXPRESS is fenestrated to help facilitate fluid movement and can be used on wounds that produce copious amounts of exudate.
  Interventions: Other: EPIXPRESS

INTERVENTIONS:
Other: Standard of Care — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Standard of Care
Other: EPIEFFECT — Participants will receive weekly applications of EPIEFFECT and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first
  Arms: EPIEFFECT
Other: EPIXPRESS — Participants will receive weekly applications of EPIXPRESS and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first
  Arms: EPIXPRESS

SUMMARY:
This study will evaluate two human amnion/chorion membrane (ppLHACM) products and Standard of Care (SOC) versus SOC alone in the closure of nonhealing diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
The CAMPAIGN trial is evaluating PURION Processed Lyophilized Human Amnion/Chorion Membrane (ppLHACM) and Standard of Care versus Standard of Care alone in the treatment of Nonhealing Diabetic Foot Ulcers. The study will evaluate two products, EPIEFFECT® and EPIXPRESS™, which are both ppLHACMs.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older.
2. Diagnosis of type 1 or 2 Diabetes mellitus.
3. At randomization subjects must have a target ulcer with a minimum surface area of 0.7 cm^2 and a maximum surface area of 5.0 cm^2 measured post debridement.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care, prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. Ankle-Brachial Index (ABI) between 0.7 and ≤ 1.3;
   2. Toe-Brachial Index (TBI) ≥ 0.6;
   3. Transcutaneous Oxygen Measurement (TCOM) ≥ 40 mmHg;
   4. Pulse Volume Resistance (PVR): biphasic.
8. If the potential subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
10. The potential subject must consent to using the prescribed offloading method for the duration of the study.
11. The potential subject must agree to attend the weekly study visits required by the protocol.
12. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. The potential subject is known to have a life expectancy of < 6 months.
2. The potential subject's target ulcer is not secondary to diabetes.
3. The target ulcer is infected or there is cellulitis in the surrounding skin.
4. The target ulcer exposes tendon or bone.
5. There is evidence of osteomyelitis complicating the target ulcer.
6. There is an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
7. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
8. The potential subject is taking hydroxyurea.
9. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
10. The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
11. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
12. The surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). MolecuLight Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
13. The surface area measurement of the Target ulcer decreases by 20% or more during the 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1 visit during which time the potential subject received SOC.
14. The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
15. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
16. The potential subject has end stage renal disease requiring dialysis.
17. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
18. A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
19. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
20. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
21. A subject has a wound with active or latent infection is excluded.
22. A subject with a disorder that would create unacceptable risk of post-operative complications is excluded.
23. A subject with a known sensitivity to aminoglycoside antibiotics is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of target ulcers achieving wound closure | 1 - 12 weeks
  The percentage of target ulcers achieving complete wound closure in 12 weeks.

SECONDARY OUTCOMES:
Percent of wound closure area | 1 - 12 weeks
  Percentage wound area reduction from treatment visit (TV)-1 to TV-13 measured weekly with digital photographic planimetry and physical examination
Adverse Events | 1 - 12 weeks
  Number of adverse events will be evaluated weekly
Change in Pain in Target Ulcer | 1 - 12 weeks
  Change in pain in the target ulcer assessed using the Pain, Enjoyment of Life and General Activity (PEG) scale
Change in Quality of Life | 1 - 12 weeks
  Change in quality-of-life using the Wound Quality of Life (wQOL) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD, Principal Investigator — SerenaGroup, Inc.; Dennis McMahon, MD, Study Director — MiMedx Group, Inc.
Locations (1):
- SerenaGroup - Monroeville, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No